CLINICAL TRIAL: NCT05507658
Title: Tislelizumab Combined With XELOX as Neoadjuvant Therapy for G/GEJ Adenocarcinoma: A Single-center, Single-arm, Phase Ⅱ Study
Brief Title: Tislelizumab Combined With XELOX as Neoadjuvant Therapy for G/GEJ Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gang Ji -1
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with XELOX (Experimental): 1. Tirelizumab 200mg, iv.gtt, D1, Q3W;
  2. Chemotherapy:
  Oxaliplatin (130 mg/m2), iv.gtt, D1, Q3W; Capecitabine (1000mg/m2), P.O.B.I.D., D1-D14, Q3W.
  Interventions: Drug: Tislelizumab combined with Oxaliplatin and Capecitabine

INTERVENTIONS:
Drug: Tislelizumab combined with Oxaliplatin and Capecitabine — Drugs:
  1. Tistelizumab 200mg, iv.gtt, D1, Q3W;
  2. Chemotherapy (XELOX) : oxaliplatin (130 mg/m2), iv.gtt, D1, Q3W; Capecitabine (1000mg/m2), P.O.B.I.D., D1-D14, Q3W.
  Neoadjuvant therapy:
  1. Tislelizumab combined with XELOX, Q3W, for 2~3 cycles;
  2. D2 radical gastrectomy after neoadjuvant therapy.
  Adjuvant therapy:
  1. From 4 to 8 weeks after surgery, the treatment dose was the same as above;
  2. Patients who achieved MPR and non-MPR on pathological evaluation were treated with tirelizumab +XELOX 3~8 cycles;
  3. Tumor evaluation performed every 3 cycles;
  4. The maximum duration of adjuvant therapy was not more than 8 cycles.

SUMMARY:
The effective treatment of G/GEJ adenocarcinoma has always been a research hotspot in academia. In recent years, mainstream studies have shown that the treatment mode of G/GEJ adenocarcinoma has changed from single surgery mode in the past, to multi-disciplinary comprehensive treatment mode for now, which is based on surgery. Several studies indicate that for most late-stage G/GEJ adenocarcinoma, the neoadjuvant treatment model can further enhance the survival rates and prognosis of patients, compared with the combination of standard radical resection and postoperative adjuvant chemotherapy. According to The Chinese Society of Clinical Oncology (CSCO): clinical guidelines for the diagnosis and treatment of gastric cancer (Wang et al , 2021), neoadjuvant therapy and adjuvant therapy are recommended for patients with G/GEJ adenocarcinoma. However, there is still a lack of unified standards and norms for precise preoperative staging of gastric cancer, applicable population of neoadjuvant along with adjuvant therapy, and the selection of treatment regimens. Therefore, this project is aimed to carry out a single-arm, open-label, phase II clinical trial to administer tirelizumab plus XELOX for neoadjuvant management of patients diagnosed with resectable gastroesophageal junction or stomach cancer, and further explore the safety and therapeutic effect of chemotherapy together with tirelizumab in the neoadjuvant period of G/GEJ adenocarcinoma, eventually, providing a new option for the neoadjuvant treatment of G/GEJ adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent;
2. Aged 18-80 (including 18 and 80), both sexes;
3. ECOG score ≤1;
4. Biopsy histologically confirmed adenocarcinoma (including Lauren grade);
5. cT3-4a N+ M0 G/GEJ adenocarcinoma confirmed by basic ultrasound gastroscopy, enhanced CT (PET/CT), MRI or diagnostic laparoscopy;

Exclusion Criteria:

1. Histological histological diagnosis of squamous cell carcinoma (adenosquamous carcinoma mainly including squamous cell carcinoma), carcinoid, undifferentiated carcinoma or other unclassified carcinoma;
2. Patients with HER2-positive status are excluded;
3. Patients with distant metastases other than primary gastric cancer (any M1 stage);
4. Patients with contraindications (laparoscopic surgery, open surgery, neoadjuvant chemotherapy);
5. Patients who can not undergo radical surgical resection (D2 radical resection);
6. Previous antitumor therapy (including chemotherapy, radiotherapy, molecular targeted therapy and hormone therapy);
7. Previously received immunological drugs such as PD-1/PD-L1, CTLA-4 or other immunological or molecular targeted therapies;
8. When virological testing prior to screening showed any of the following:

   1. patients with active hepatitis (HBV DNA≥1*103 copies or ≥200IU/mL);
   2. Anti - HCV positive;
   3. HIV positive;
9. Patients or their families refused to sign this informed consent form to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Major pathological response rate(MPR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 years
  Defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time.

SECONDARY OUTCOMES:
Pathological complete response rate(pCR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Pathological complete response
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
TRAEs and postoperative complications | Investigator assessment,from the initiation date of the operation day, assessed up to 1 years.
  Including TRAEs and postoperative complications Complications refer to the occurrence of another or several diseases related to the therapeutic behavior of this disease during the treatment of a certain disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China